CLINICAL TRIAL: NCT05741931
Title: Monitoring Pregnant Women Using REST Mobile Application (Risk Identification, Evaluation Counseling, Systematic Monitoring, Troubleshooting)
Brief Title: Pregnancy Monitoring Using Mobile Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Restu Pangestuti, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 485838
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Maternal and Child Health
Keywords: pregnancy monitoring; mobile application; antenatal care; maternal and child health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Pregnant women and midwives will use the REST (Risk identification, Evaluation counseling, Systematic monitoring, Troubleshooting) mobile application to monitor the condition of maternal pregnancy. Mothers and midwives will implementation 3 times of pregnancy class until mothers give birth
  Interventions: Device: mobile application REST (Risk identification, Evaluation counseling, Systematic monitoring, Troubleshooting)
- Control Group (No Intervention): Pregnant women and midwives will conduct pregnancy monitoring as usual. The pregnancy class will be implemented in accordance with government program standards. Mothers will take pregnancy class 3 times until the mother gives birth

INTERVENTIONS:
Device: mobile application REST (Risk identification, Evaluation counseling, Systematic monitoring, Troubleshooting) — The mobile application will be installed on the mobile phone. The application is used to monitor pregnant women. Users of the application are midwives and pregnant women. The application contains documentation of the health condition of pregnant women.
  Arms: Intervention Group

SUMMARY:
The goal of this Randomized Controlled Trial is to compare the health condition of pregnant women through pregnancy monitoring in the implementation of pregnancy class. The main question it aims to answer are:

How is the condition of the mother and baby after pregnancy monitoring using the REST mobile application (Risk identification, Evaluation counseling, Systematic monitoring, Trobleshooting)

Participants will be monitored for the condition of their pregnancy from 20 weeks of pregnancy until delivery. Participants will attend in the pregnancy class as many as 3 meetings and a pregnancy check-up by the midwife.

Researchers will compare intervention group to see if normal delivery methods, birth weight of the baby (>2500), antenatal care visits (>6 times), and prevention of pregnancy complications were better than the control group.

DETAILED DESCRIPTION:
The research will involve pregnant women and midwives. The midwife will conduct a pregnancy check-up which includes 10 pregnancy checks (height and weight, blood pressure, upper arm circumference, uterine fundus height, Tetanus immunization, Fe tablets, fetal presentation and fetal heart rate, counseling, laboratory tests, case handling). The examination is carried out every class meeting of pregnant women. The results of the examination will be inputted into the mobile application. Pregnant women will fill in the mobile application if the mother does antenatal care at a health facility. This activity will last until the mother's delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a gestational age of 20-22 weeks.
* Pregnant women who have a pregnancy check-up at a health facility
* Plan to settle in the research area for at least the next 2 years
* Willing to participate in the research by signing an informed consent form.

Exclusion Criteria:

* Suffering from chronic diseases that require special pregnancy care
* It is certain that it cannot give birth normally
* Unable to operate an android phone

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 216 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Reduced incidence of pregnancy complications in the mother | 20 weeks gestational age until delivery
  Pregnancy complications are measured using a mobile application by looking at the history of the mother's health condition. Possible complications such as pre-eclampsia, eclampsia, hypertension in pregnancy, and anemia
Increased childbirth by normal methods | 20 weeks gestational age until delivery
  The delivery method can be seen using the mobile application in the labor report section. Delivery will be reported by the midwife regarding the method used for childbirth including the results of filling out the partograph
Reduced incidence of low birth weight babies | 20 weeks gestational age until delivery
  The baby's birth weight is measured using baby scales and it is expected that the baby's birth weight is more than 2500 grams
Antenatal care for pregnant women more than 6 visits | During pregnancy
  Antenatal care by mothers can be measured by the number of visits to health facilities for pregnancy check-ups. Each visit will be recorded on the mobile application starting from the first visit

CONTACTS AND LOCATIONS:
Overall Officials: Prima D Ratrikaningtyas, Study Chair — Gadjah Mada University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pangestuti R, Ratrikaningtyas PD, Sutomo AH. Monitoring of Pregnant Women Using the "Risk Identification, Evaluation Counseling, Systematic Monitoring, Troubleshooting" (REST) Mobile App: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 6;14:e66774. doi: 10.2196/66774. PMID 40768267